CLINICAL TRIAL: NCT06014294
Title: Effects of High-Intensity Interval Training on Depressive Symptoms in Hong Kong Older Adults With Mild and Moderate Depression: A Cluster-Randomized Controlled Trial
Brief Title: Effects of High-Intensity Interval Training on Depressive Symptoms in Hong Kong Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12616922
Record Dates: First submitted 2023-08-08; First posted 2023-08-28 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-06

CONDITIONS: Depressive Symptoms
Keywords: Depressive symptoms; Older adults; High-intensity interval training; Baduanjin Qigong
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The present research follows a cluster randomized controlled experimental design (CRCT), parallel type with three groups in multi-centers and being assessed in a pretest, posttest, and after three months of the completion of the intervention. The participants will be randomly allocated to one experimental group, one exercise control group, and one non-exercise control group. The non-exercise control group continue to maintain their daily routine and will be asked to attend workshop. While two exercise groups, one group performs a HIIT program, and the other group performs a Baduanjin exercise program.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (HIIT) (Experimental): HIIT program for 16 weeks with a frequency of 2 times per week.
  Interventions: Behavioral: HIIT
- Moderate intensity continuous training (MICT) (Active Comparator): Baduanjin exercise as MICT will be applied with the same program duration and frequency as the HIIT group. The entire set of Baduanjin Qigong exercises in the current study includes 8 postures.
  Interventions: Behavioral: Baduanjin
- Non-exercise control (Placebo Comparator): Participants will not receive any exercise training, but attending 32 recreation workshops.
  Interventions: Behavioral: Workshop

INTERVENTIONS:
Behavioral: HIIT — Participants will receive a 16-week HIIT program, with 2 sessions per week. Each session will comprise three sections, including warm-up, main exercise and cool down. The time will be between 34 to 40 minutes with progression of training. Each HIIT section will include ten combined exercises with self-weight. For Weeks 1-2, the HIIT section will include 10 intervals of 30 seconds HIIT workout at corresponding intensity, separated by 9 intervals of 60 seconds of active recovery.
  Arms: High-intensity interval training (HIIT)
Behavioral: Baduanjin — As a typical MICT, Baduanjin Qigong will be performed. The instructor will provide group teaching with individual instructions on specific movements. The same training principles of individuality and progression used in the HIIT group will also be applied to Baduanjin Qigong group.
  Arms: Moderate intensity continuous training (MICT)
Behavioral: Workshop — Participants in the non-exercise control group will receive a series of workshops related to daily recreation.
  Arms: Non-exercise control

SUMMARY:
Depression in later life is a common health problem in aging societies. It is associated with poor quality of life, and increased risks of morbidity and mortality. People with severe depression may develop serious psychotic symptoms (e.g., delusions) and have higher mortality and disability than those with mild and moderate depression.

Traditional moderate-intensity continuous training (MICT) (e.g., Baduanjin Qigong) has proved to be effective in preventing and alleviating depressive symptoms among older adults. However, older adults with mental illnesses have poorer engagement and compliance with MICT programs. In recent years, as a novel type of exercise, high-intensity interval training (HIIT), which includes repeated bouts of high-intensity effort followed by varied recovery times, appears to be a promising approach for overcoming limitations in traditional MICT programs.

Considering there is little evidence of HIIT benefits related to older adults with depression, the current study aims to evaluate the effectiveness of a 16-week HIIT intervention on depressive symptoms and other health-related outcomes among Hong Kong Chinese older adults.

DETAILED DESCRIPTION:
The study will be a cluster randomized controlled trial (CRCT) with three groups and three times repeated measures. Data will be collected in a pretest, post-test, and three months after the intervention. The eligible community elderly centers will be randomly distributed into one of three groups in a ratio of 1:1:1. The participants recruited and meeting the screening criteria will receive a 16-week HIIT intervention or Baduanjin exercise or recreation workshop. The intervention effects will be evaluated on depressive symptoms, concentration of salivary cortisol, sleep quality, quality of life, and physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 74 years at the start date of the project
* Chinese version of Geriatric Depression Scale (GDS-C) scoring 5-11 (i.e., mild to moderate level of depressive symptoms)
* Passing the PAR-Q plus screening or with the physician's approval for readiness to participate in high-intensity exercise
* Above the average level of 2-mins stepping showing competent aerobic fitness
* No restriction on physical mobility
* No cognitive impairment, as determined by the Chinese version of the Mini-Mental Status Examination (i.e., score < 24)
* No previous substantial experiences in practicing HIIT or Baduanjin Qigong. The written informed consent form will be collected from each participant

Exclusion Criteria:

* Severe chronic disease restricting high-intensity exercise
* Having cognition impairment regarded by specialists

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported depressive symptoms | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  The Chinese version of the 15-item Geriatric Depression Scale (GDS-C) will be used to measure the subjective depression level. The GDS are the most widely used scales for the detection of depression symptoms in older adults (Cronbach's α = .81 -.83).

SECONDARY OUTCOMES:
Concentration of saliva cortisol | Evaluations of concentration of saliva cortisol will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  Objective biomarker of depression will be measured in salivary cortisol. All participants will be provided with three salivette tubes and be asked to collect the saliva samples (2-3 ml) at awakening and 30 mins after awakening, respectively. All saliva samples for all subjects will be collected at the same time of day and samples will not be taken on days in which participants are sick with a fever. The salivette tubes will be stored in the freezer zone until to be tested. ELISA KIT protocol will be used to be followed to collect and analyze the samples in each assessment.
Physical fitness | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  Physical fitness will be assessed using the Senior Fitness Test (SFT) battery. There are seven testing items measuring all five dimensions of PT, including the body mass index (BMI), 30s chair stand for lower limbs' muscle strength, 30s arm curl for upper limbs' muscle strength, 2-min step test for aerobic endurance, chair sit-and-reach test for lower body flexibility, back scratch test for upper body flexibility, and 8ft up-and-go test for mobility and dynamic balance.
Sleep quality | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  The Chinese version of the Pittsburgh Sleep Quality Index (PSQI) will be used to measure sleep quality. The PSQI is a widely validated scale appropriate for use with older adults. The scale includes 18 items, covering seven domains: subjective SQ, sleep latency, sleep duration, sleep efficiency, frequency of sleep disturbance, daytime dysfunction, and use of sleep medications.
Perceived quality of life | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  The quality of life will be assessed by the Hong Kong Chinese WHO Quality of Life Scale brief version (WHOQOL-BREF) (Cronbach's α = .73 -.84). The scale includes 28 items, covering four dimensions of how older adults perceive their quality of life.

OTHER OUTCOMES:
Heart rate | Heart rate will be monitored from the start of warm-up to the end of cool-down at each exercise session during the 16-weeks exercise intervention.
  Participants will be monitored by Polar verity sensor during exercise and their heart rate will be monitored to ensure their safety and intensity adherence of exercise protocol.
Self-reported Rate of Perceived Exertion (RPE) | RPE will be asked at the end of main exercise at each exercise session during the 16-weeks intervention.
  Older adults will be asked about the self-reported Rate of Perceived Exertion (RPE Borg CR-10 category scale) after they complete the main exercise training in each session.
Safety: adverse events | Adverse events will be asked at the end of each exercise session during the 16-weeks intervention program.
  All adverse events will be recorded as safety endpoints.
Exercise acceptability | Outcome evaluations will be conducted at the completion of 16-weeks intervention.
  Exercise acceptability will be assessed post-intervention using ten questionnaire items responding to a 5-point Likert scale (strongly disagree, disagree, neither agree nor disagree, agree, and strongly agree). The score on this scale ranges from 10 to 50, the higher score shows better acceptability to the exercise intervention.
Process evaluation of intervention program | Outcome evaluations will be conducted at the completion of 16-weeks intervention.
  A process evaluation scale of the intervention process will be developed for this study based on the previous framework of process evaluation for the intervention study. This scale with 10 items using a 5-point (strongly unsatisfied, unsatisfied, neutral, satisfied, and strongly satisfied). The score on this scale ranges from 10 to 50, a higher score shows higher satisfaction with the intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Duan, Principal Investigator — Hong Kong Baptist Univeristy; Department of Sport, Physical Education and Health
Locations (1):
- Bliss District Elderly Community Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung GT, de Jong Gierveld J, Lam LC. Validation of the Chinese translation of the 6-item De Jong Gierveld Loneliness Scale in elderly Chinese. Int Psychogeriatr. 2008 Dec;20(6):1262-72. doi: 10.1017/S1041610208007552. Epub 2008 Jul 1. PMID 18590603
- [Background] Wei J, Hou R, Zhang X, Xu H, Xie L, Chandrasekar EK, Ying M, Goodman M. The association of late-life depression with all-cause and cardiovascular mortality among community-dwelling older adults: systematic review and meta-analysis. Br J Psychiatry. 2019 Aug;215(2):449-455. doi: 10.1192/bjp.2019.74. Epub 2019 Apr 10. PMID 30968781
- [Background] Liu F, Cui J, Liu X, Chen KW, Chen X, Li R. The effect of tai chi and Qigong exercise on depression and anxiety of individuals with substance use disorders: a systematic review and meta-analysis. BMC Complement Med Ther. 2020 May 29;20(1):161. doi: 10.1186/s12906-020-02967-8. PMID 32471415
- [Background] Zou L, Pan Z, Yeung A, Talwar S, Wang C, Liu Y, Shu Y, Chen X, Thomas GA. A Review Study on the Beneficial Effects of Baduanjin. J Altern Complement Med. 2018 Apr;24(4):324-335. doi: 10.1089/acm.2017.0241. Epub 2017 Dec 11. PMID 29227709
- [Background] Martland R, Mondelli V, Gaughran F, Stubbs B. Can high intensity interval training improve health outcomes among people with mental illness? A systematic review and preliminary meta-analysis of intervention studies across a range of mental illnesses. J Affect Disord. 2020 Feb 15;263:629-660. doi: 10.1016/j.jad.2019.11.039. Epub 2019 Nov 12. PMID 31780128
- [Background] Martland R, Korman N, Firth J, Vancampfort D, Thompson T, Stubbs B. Can high-intensity interval training improve mental health outcomes in the general population and those with physical illnesses? A systematic review and meta-analysis. Br J Sports Med. 2022 Mar;56(5):279-291. doi: 10.1136/bjsports-2021-103984. Epub 2021 Sep 16. PMID 34531186
- [Background] Korman N, Armour M, Chapman J, Rosenbaum S, Kisely S, Suetani S, Firth J, Siskind D. High Intensity Interval training (HIIT) for people with severe mental illness: A systematic review & meta-analysis of intervention studies- considering diverse approaches for mental and physical recovery. Psychiatry Res. 2020 Feb;284:112601. doi: 10.1016/j.psychres.2019.112601. Epub 2019 Nov 28. PMID 31883740
- [Background] Cheng ST, Chan AC. A brief version of the geriatric depression scale for the chinese. Psychol Assess. 2004 Jun;16(2):182-6. doi: 10.1037/1040-3590.16.2.182. PMID 15222814
- [Background] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Background] Rikli RE, Jones CJ. Senior fitness test manual. Human kinetics; 2013
- [Background] Chen HC, Hsu NW, Chou P. Subgrouping Poor Sleep Quality in Community-Dwelling Older Adults with Latent Class Analysis - The Yilan Study, Taiwan. Sci Rep. 2020 Mar 25;10(1):5432. doi: 10.1038/s41598-020-62374-4. PMID 32214167
- [Background] Leung KF, Tay M, Cheng SS, Lin F. Hong Kong Chinese version World Health Organization quality of life measure-abbreviated version. Hong Kong: Hong Kong Hospital Authority. 1997 Dec.
- [Background] Chapman, J. J., Coombes, J. S., Brown, W. J., Khan, A., Chamoli, S., Pachana, N. A., & Burton, N. W. (2017). The feasibility and acceptability of high-intensity interval training for adults with mental illness: A pilot study. Mental Health and Physical Activity, 13, 40-48.
- [Background] Grant A, Treweek S, Dreischulte T, Foy R, Guthrie B. Process evaluations for cluster-randomised trials of complex interventions: a proposed framework for design and reporting. Trials. 2013 Jan 12;14:15. doi: 10.1186/1745-6215-14-15. PMID 23311722
- [Derived] Duan Y, Wang Y, Liang W, Wong HS, Baker JS, Yang S. Feasibility and effects of high-intensity interval training in older adults with mild to moderate depressive symptoms: A pilot cluster-randomized controlled trial. J Exerc Sci Fit. 2025 Jul;23(3):246-251. doi: 10.1016/j.jesf.2025.05.004. Epub 2025 May 24. PMID 40520628
- See also: World Health Organization. Depression (2020). — https://www.who.int/news-room/fact-sheets/detail/depression
- See also: Non-Communicable Diseases Watch. (2012). Depression: Beyond Feeling Blue. — https://www.chp.gov.hk/files/pdf/ncd_watch_sep2012.pdf